CLINICAL TRIAL: NCT02940561
Title: A Multicenter, Randomized, Open Label, Two Treatment, Two Period, Two Sequence, Single-dose, Two-way, Crossover, Bioequivalence Study of Methotrexate Tablets USP, 2.5 mg Manufactured by Amneal Pharmaceuticals, With Methotrexate Tablets USP 2.5 mg Manufactured for DAVA Pharmaceuticals, Inc., Fort Lee, NJ 07024 USA in Patients With Mild to Severe Psoriasis or Rheumatoid Arthritis, Who Are Already on Established Regimens of 2.5 mg Every 12 Hours Under Fasting Condition.
Brief Title: BE Study in Patients - Methotrexate Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amneal Pharmaceuticals, LLC (Industry)
Collaborators: Accutest Research Laboratories (I) Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 15-VIN-515
Record Dates: First submitted 2016-09-15; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Psoriasis; Rheumatoid Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate - Amneal (Experimental): Methotrexate Tablets USP, 2.5 mg, single-dose in each period
  Interventions: Drug: Methotrexate - Amneal
- Methotrexate - DAVA (Active Comparator): Methotrexate Tablets USP, 2.5 mg, single-dose in each period
  Interventions: Drug: Methotrexate - DAVA

INTERVENTIONS:
Drug: Methotrexate - Amneal — Methotrexate Tablets, USP contain an amount of methotrexate sodium equivalent to 2.5 mg of methotrexate, USP and are round, biconvex, yellow tablets, scored in half on one side, engraved with "A" above the score and "1" below
  Other Names: Methotrexate Sodium
  Arms: Methotrexate - Amneal
Drug: Methotrexate - DAVA — Methotrexate Tablets, USP contain an amount of methotrexate sodium equivalent to 2.5 mg of methotrexate and are round, convex, yellow tablets, scored in half on one side, engraved with M above the score, and 1 below
  Other Names: Methotrexate Sodium
  Arms: Methotrexate - DAVA

SUMMARY:
To characterize the pharmacokinetic profile of the Test product - Methotrexate Tablets USP, 2.5 mg of Amneal Pharmaceuticals, compared to that of the corresponding Reference product - Methotrexate Tablets USP 2.5 mg manufactured for DAVA Pharmaceuticals, Inc. in patients with mild to severe psoriasis or rheumatoid arthritis, who are already on established regimens of 2.5 mg every 12 hours for three doses per week under fasting conditions, and to assess their bioequivalence.

DETAILED DESCRIPTION:
Patients will continue their own established dose of 2.5 mg tablet at 12 hours intervals for 3 doses given as a course once weekly. This dosing regimen will be kept constant throughout the study period.

On day 0 of each period, the patient will be hospitalized/ housed in the clinical facility/hospital, so patient will be administered IP dose on day 1 under supervision of trained study staff.

In supervised dosing, patient will be administered oral dose of Methotrexate Tablet 2.5 mg (Test or Reference product as per randomization schedule) with approximately 240 mL of water at ambient temperature in sitting position. Mouth check will be done by investigator/ designee followed by IP administration to verify dosing compliance.

The patient will be advised to take two subsequent doses of the locally approved drug at every 12 hours of interval after the administration of study drug on day 1.

Compliance to subsequent two doses of locally approved Methotrexate tablets 2.5 mg will be ensured as below in each period.

The dose which is to be given 12 hours after IP administration (Second dose) will be administered inside clinical facility after collection of 12 hours post-dose PK sample under supervision of trained study personnel. The next dose (third dose) will be provided to the patients with the instruction to take the same on their own. Telephonic follow-up will be made on the next day for this third dose. The same will be documented in the patient dosing log.

In period I, patient will be housed on day 0 at least 12 hours prior to IP dosing scheduled on day 1 and will remain in clinical facility till last PK sample on day 1. Patient will be checked out on day 1 after last PK blood sample collection followed by administration of second dose of locally approved Methotrexate 2.5 mg tablet. The third dose of locally approved Methotrexate 2.5 mg tablet should be taken by patient on their own approximately 12 hours after the second dose.

The same procedure will be followed in period II.

There will be a period of at least 7 days between first dosing (IP administration) in both the study periods.

The patients will have to stay hospitalized for a period of 2 days and 1 night in each study period for their convenience and close safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to severe psoriasis or rheumatoid arthritis, who are already on established regimens of 2.5 mg every 12 hours (7.5 mg per week in three divided doses)
* Confirmed diagnosis of psoriasis by clinical examination or after dermatologic consultation.

or confirmed diagnosis of mild to severe rheumatoidarthritis based on at least 1 of the following: i. Documented history of positive rheumatoid factor ii. Current presence of rheumatoid factor iii. Radiographic erosion within 12 months prior to enrollment iv. Presence of serum anti-cyclic citrullinated peptide antibodies (anti-CCP).

* Women of childbearing potential (include girls who have entered puberty and all women who have a uterus and ovaries and have not completed menopause wherein menopause is the permanent end of menstruation and fertility. Females who have 12 consecutive months of spontaneous amenorrhea (not induced by a medical condition or medical therapy) or have bilateral absence of ovaries (surgical or congenital) have completed menopause must have a negative serum pregnancy test at screening and negative urine pregnancy test on check in to housing, and must agree to use an adequate method of contraception.
* Patient's screening laboratory assessment (complete blood count [CBC] and blood chemistries) are clinically non-significant as per the discretion of the Investigator.
* No history of addiction to any recreational drug or drug dependence.
* No participation in any clinical study within the past 60 days prior to receiving the first dose of investigational product for the current study.

Exclusion Criteria:

* A history of allergic or adverse reactions to Methotrexate Sodium or any related drug or any excipient of methotrexate tablets.
* Females of childbearing potential unwilling to use adequate contraception (as defined in the protocol) throughout the trial and for one month after the last dose of study medication.
* Males unwilling to use a male condom throughout the trial and for three months after the last dose of study medication
* Patients with alcoholism, alcoholic liver disease or other chronic liver disease.
* Patients who are diagnosed to be HIV or Hepatitis B (HBsAg) or Hepatitis C (HCV) virus reactive/positive.
* Patients who have clinically significant abnormal laboratory values at screening.
* Patients with any evidence of organ dysfunction or any clinically significant deviation from normal in their physical or clinical evaluation including ECG and X-ray results except study indication.
* Patients who have overt or laboratory evidence of immunodeficiency syndromes.
* Patients currently suffering from or having a history of malignant lymphoma or tumor lysis syndrome.
* Patients who have pre-existing hematopoietic impairment/ blood dyscrasias, such as bone marrow hypoplasia, aplastic anemia, pancytopenia, leukopenia, neutropenia, thrombocytopenia and or significant anemia.
* Patient with lymphadenopathy and lymphoproliferative disorders.
* Patients suffering from any acute infection within two weeks prior to randomization.
* Patients with a clinically significant past history or current medical condition of: Pulmonary disorders (Pneumonia, COPD and asthma), pleural effusions, Cardiovascular disorders (especially cardiac blocks, pericarditis, pericardial effusion, hypotension and thromboembolic events ), Neurological disorders (especially seizures, migraines), Gastrointestinal tract disorders including a history or presence of significant gastric and/or duodenal ulceration and bleeding, hematemesis, melena, enteritis, pancreatitis, Renal and/or hepatic disorders, Coagulation disorders, Patient with ascites, Patient with uncontrolled diabetes mellitus.
* Female patients who are pregnant or breastfeeding
* History or presence of cancer.
* Evidence of any significant uncontrolled concomitant disease which in the investigator's opinion would exclude the patient participation.
* Expected changes in concomitant medications during the period of study.
* Tested positive for Alcohol breath or Urine drug of abuse.
* Any treatment which could affect the pharmacokinetic of methotrexate (NSAIDs, salicylates, hypoglycemics, diuretics, sulphonamides, diphenylhydantoins, tetracyclines, chloramphenicol and p-aminobenzoic acid, probenecid, penicillins, Chloroquine, omeprazole, etretinate, co-trimoxazole and trimethoprim etc.) administered within 1 month of starting of study.
* Patient had major surgery within 4 weeks prior to study entry, or who have not recovered from prior major surgery.
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
* History of difficulty with donating blood or difficulty in accessibility of veins.
* Patients for whom oral administration of drug is not possible.
* An unusual or abnormal diet, for whatever reason e.g. religious fasting.
* Blood donation/ loss exceeding 200 ml within last 60 days prior to receiving the first dose of investigational product for the current study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC0-12) | Blood samples will be collected on day 1 of each period, pre-dose and post-dose at 0.167, 0.333, 0.500, 0.750, 1.000, 1.250, 1.500, 1.750, 2.000, 2.333, 2.667, 3.000, 3.500, and 4 hours
  The area under the plasma concentration versus time curve, from time 0 to 12 hours post-dose, calculated using linear trapezoidal method. It will be calculated using plasma concentration vs. time profile (Actual time of sample collection) data of the investigational products in individual subjects.
Maximum Plasma Concentration (Cmax) | Blood samples will be collected on day 1 of each period, pre-dose and post-dose at 0.167, 0.333, 0.500, 0.750, 1.000, 1.250, 1.500, 1.750, 2.000, 2.333, 2.667, 3.000, 3.500 and 4 hours
  Maximum measured plasma concentration over the time span specified. It will be calculated using plasma concentration vs. time profile (Actual time of sample collection) data of the investigational products in individual subjects.

SECONDARY OUTCOMES:
Safety Parameters | through study completion, approximately 23 days
  Safety parameters will include monitoring of AEs, SAEs, physical examination results, vital signs and clinical laboratory results

CONTACTS AND LOCATIONS:
Overall Officials: Prayag N Shah, MD, Study Director — Amneal Pharmaceuticals
Locations (3):
- India (3):
  - Saviour Hospital, Ahmedabad, Gujarat
  - Sterling Hospital, Ahmedabad, Gujarat
  - Kanoria Hospital, Gandhinagar, Gujurat

IPD SHARING:
Plan to Share IPD: No